CLINICAL TRIAL: NCT07289360
Title: Testing a Mixed-Reality Video Game for Home-Based Practice of Arm-Hand Skills for Children With Cerebral Palsy: A Pilot Randomized Controlled Trial
Brief Title: Bootle Blast: Pilot Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Elaine Biddiss, Principal Investigator, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1954
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Hemiplegic Cerebral Palsy
Keywords: Home-Based Rehabilitation; Interactive Video Game Therapy; Digital Therapeutics; Tele-Rehabilitation; Gamified Rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a 24-week mixed-methods pilot randomized controlled trial using a parallel-group design. Participants are allocated by minimization to either the Experimental Group, which receives the Bootle Blast intervention immediately, or the Waitlist Comparison Group, which continues standard care for the first 12 weeks. Both groups complete in-person assessments at 0, 12, and 24 weeks. After the 12-week assessment, the Waitlist Group receives the same Bootle Blast intervention. Within each arm, participants are further randomized to receive or not receive weekly monitoring coach calls to explore added support effects. Repeated measurements (system logs, clinical assessments, COPM-goal videos, and engagement metrics) are collected throughout to evaluate the feasibility and acceptability of conducting a larger-scale RCT.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Occupational therapists administering the clinical assessments at 0, 12, and 24 weeks are blinded to group allocation. All assessments are video recorded and subsequently scored, with some scored by separate blinded raters who are also unaware of group assignment and time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bootle Blast Play Phase (0 - 12 weeks) followed by Standard Care (12 - 24 weeks) (Experimental): Participants receive the Bootle Blast home-based intervention immediately after baseline in-person clinic assessment at 0 weeks. Families complete 12 weeks of home-based play targeting a prescribed practice dose (15-20 minutes/day, 3-4 days/week), alongside ongoing standard care activities. Participants may also be randomized to receive weekly monitoring coach calls providing motivational and technical support. Participants complete in-person clinical assessments again at 12 and 24 weeks, and provide repeated COPM-goal videos, PRIME engagement data, and system-logged play data during the intervention period. After the 12-week assessment, they transition to standard care without Bootle Blast for weeks 12-24.
  Interventions: Device: Bootle Blast Intervention; Other: Standard Care (Comparator)
- Waitlist Comparison - Standard Care (0-12 weeks) followed by Bootle Blast Play Phase (12-24 weeks) (Other): Participants continue with their usual standard care for the first 12 weeks after baseline assessment. During this period, they do not receive Bootle Blast but complete the same assessment schedule and repeated measures as the experimental group. After the 12-week assessment, they receive the Bootle Blast intervention following the same calibration and training procedure, with randomized monitoring coach support. They then complete the 12-week Bootle Blast period from weeks 12 to 24, along with follow-up assessments and repeated measurements. This group is likely representative of how Bootle Blast would be used in practice (complement or supplement to standard care).
  Interventions: Device: Bootle Blast Intervention; Other: Standard Care (Comparator)

INTERVENTIONS:
Device: Bootle Blast Intervention — Bootle Blast is a movement-tracking, mixed-reality therapeutic video game delivered in the home using the Orbbec Persee 3D camera-computer. An occupational therapist calibrates the system to each child's range and speed of motion and targeted therapy goals. Families are trained to set up and use the system. Participants then complete 12 weeks of home-based practice targeting 15-20 minutes per day, 3-4 days per week. The system automatically records active play time, movement counts, and performance data. Some participants are randomized to receive weekly monitoring coach phone calls for motivational and technical support.
Other: Standard Care (Comparator) — Participants continue with their usual care, which may include routine stretching, maintenance exercises, and consultative visits with their healthcare professionals. Targeted upper-limb therapies (e.g., constraint therapy, botulinum toxin, casting) are excluded during the study period.

SUMMARY:
One in 500 Canadians has cerebral palsy (CP), a lifelong condition affecting movement and function. Physical and occupational therapies greatly benefit children with CP but can be costly and difficult to access. Children, parents, and clinicians are interested in using movement-tracking video games for home-based hand/arm therapy. Yet, the technologies and evidence to support this approach are limited. We partnered with key stakeholders and an interdisciplinary team to co-create Bootle Blast. Bootle Blast tracks skeletal movements and interactions with real-life objects, engaging children in individualized play experiences rich in feedback, task specificity, and opportunities for goal-directed motor practice linked to meaningful activities.

To establish Bootle Blast's clinical effectiveness, a large-scale randomized controlled trial (RCT) is needed. Pilot RCTs provide important insights that position large-scale RCTs for success. As a result, the goal of this Pilot RCT is to test whether a mixed-reality video game intervention (i.e. Bootle Blast) can improve upper-limb function, activity, and participation in children and youth aged 6-17 years with hemiplegic cerebral palsy. The main questions it aims to answer are: (1) Is it feasible and acceptable for families to use Bootle Blast at home for 12 weeks? (2) Does the intervention show preliminary improvements in hand-arm motor outcomes compared to usual care?

Researchers will compare an immediate Bootle Blast intervention group to a waitlist comparison group that continues usual care for 12 weeks to see whether access to Bootle Blast leads to increased practice, greater engagement, and improved motor outcomes.

Participants will:

Complete three in-person assessments (baseline, 12 weeks, 24 weeks) with standardized motor and participation measures.

Be randomized to begin 12 weeks of home-based Bootle Blast immediately or after a 12-week waitlist period.

Use the Bootle Blast game at home for 15-20 minutes per day, 3-4 days per week, with all gameplay tracked automatically.

A subset of participants will also receive weekly 10-minute support calls from a monitoring coach.

DETAILED DESCRIPTION:
One in 500 Canadians has cerebral palsy (CP), a lifelong condition affecting movement and function.CP is the most common cause of physical disability in children. Hemiplegic CP (~40% of CP diagnoses) affects one side of the body impacting arm/hand function. Between 60% and 83% of children with CP have upper limb involvement that can impact independence in activities of daily living, school and leisure, and social participation. Occupational and physiotherapy can help improve and/or maintain the many components of arm and hand function including gripping/releasing objects, reach, speed and accuracy, grip strength, and sensibility, often mitigating need for surgical interventions. While benefits of therapy can be significant, costs to the healthcare system and families are rising. Costs to manage CP over a lifetime average $1.2 million/person. Demand for therapy outpaces availability. In rural areas, families travel far to access services. While home-based therapy can improve outcomes, nearly half of families report low adherence due to limited time, lack of motivation, or forgetfulness. Sustaining child and parent motivation in home-based motor therapies is a long-standing challenge of great importance in pediatric practice. In fact, clinicians rate child motivation to be the most influential trait predicting success in motor therapies for CP. There is a clear need for new approaches to motivate and support children and families in home-based therapy.

In line with this need, families and clinicians at Holland Bloorview Kids Rehabilitation Hospital (Holland Bloorview) and partner organizations affiliated with Empowered Kids Ontario (EKO), asked: can we use video games to create fun, effective opportunities for motor practice for children with CP? Finding no suitable video games to support hand/arm therapy, we partnered with diverse knowledge users (i.e. children with CP, their siblings, caregivers, clinicians), interdisciplinary researchers, specialists (e.g. engineers, games developers) and with guidance from provincial networks (CP-Net) and external partnerships (MaRS Innovation; Ubisoft), developed Bootle Blast. Bootle Blast was designed to overcome established limitations of video games currently used for hand-arm therapy including: lack of feedback, inability to target specific therapy goals and/or sustain engagement, and solo gameplay. Bootle Blast is the first video game for hand-arm therapy that systematically integrates best practices in motor learning, motivational theory, and game design. Using the Orbbec Persee (a 3D camera-computer), Bootle Blast provides real-time feedback on skeletal movements and interactions with real-life objects used in gameplay (e.g. building blocks) that is tracked over time. This "mixed reality" play experience offers greater task specificity to enhance transfer of skills to everyday activities. It enables individualized treatment plans by supporting practice of a wide range of motor skills with activities that can be calibrated to each child's abilities. Bootle Blast enables people of different abilities to play meaningfully together, enhancing social equalization. Game rewards are directly linked to therapeutic effort and incentivize frequent practice of goal-directed movements. These 5 attributes (feedback, task specificity, individualized treatment plans, social equalization, practice) are considered the system-level "active ingredients" of interactive computer play for motor learning, while therapist support is considered an intervention-level "active ingredient" that can impact participant motivation and outcomes. Bootle Blast is the first technology to deliver all five active ingredients, while also applying engaging game design principles. With support from CIHR, NSERC and the Ontario Brain Institute, Bootle Blast has been iteratively co-created and tested with the Children's Advisory Council, in clinics, and with research participants culminating in a refined technology that reflects the lived experiences of our knowledge users.

To establish the clinical effectiveness of Bootle Blast, a well-designed randomized controlled trial (RCT) is now needed. Efficacy RCTs are resource intensive. Pilot RCTs provide critical insights that position efficacy RCTs for success and help to ensure that resources are invested in trials likely to generate clinically meaningful results.

Consequently, this pilot randomized controlled trial will examine whether it is feasible and acceptable to conduct a larger RCT to determine whether 12 weeks of home-based Bootle Blast use can improve upper-limb function, activity, and participation outcomes in children with hemiplegic CP compared to standard care. The study uses a mixed-methods design with a waitlist comparison group. Children aged 6-17 years with hemiplegic CP (MACS I-III) will be randomized using minimization to balance age, sex, and MACS level. The intervention group will receive Bootle Blast immediately for 12 weeks, while the comparison group continues their usual care for 12 weeks before crossing over. A subset of participants in each arm will be randomly assigned to receive weekly support from a monitoring coach to investigate whether coach contact affects adherence, engagement, or outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegic Cerebral Palsy
* MACS levels I (handles objects easily) to III (handles objects with difficulty)
* Aged 6 to 17 years with sufficient cognitive capacity and cooperation to play Bootle Blast and complete outcome assessments
* Ability to communicate in English
* Able to travel to Holland Bloorview, Grandview or CHEO and complete a total of 3 in-person study appointments
* Has a large screen (e.g. TV) with an appropriate play space (3m x 3m) in front
* At least intermittent access to the internet
* Have time to play Bootle Blast for 15-20 minutes/day, 3-4 days/week for 12 weeks.

Exclusion Criteria:

* Received upper limb surgery, botulin toxin injections in the past 4 months, or constraint therapy/casting in the previous 3 months that may be associated with changing abilities
* Currently or anticipates receiving active treatments impacting upper limb function during the study period
* Uncontrolled epilepsy that may be triggered by video game play
* Medical condition impeding safe participation in physical activity associated with Bootle Blast
* Visual limitations that interfere with Bootle Blast play

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Throughout 24-week study period.
  Number of participants enrolled per month across all study sites. Assessed against feasibility criterion of ≥4 participants/month.
Attrition Rate | Throughout 24-week study period.
  Number and proportion of enrolled participants who do not complete the scheduled assessments at 12 or 24 weeks. Feasibility criterion: <15% attrition.
Adherence to Bootle Blast Intervention | Weeks 0-12 (Experimental Group), Weeks 12-24 (Waitlist Comparison Group).
  Adherence measured using system-logged data, including minutes of active therapeutic play, passive play, and number of intentional therapeutic movements (e.g., reach, cross-body reach, grasp-and-release). Target dose: ≥10 hours of active play over 12 weeks.
Intervention Acceptability Survey | Week 12 (Experimental Group), Week 24 (Waitlist Comparison Group).
  Child and parent ratings of (i) satisfaction with the Bootle Blast intervention (e.g. therapeutic content, game content, challenge level, support provided), (ii) perceived impact and any unmet needs; and (iii) appropriateness and burden of study protocols (e.g. outcome measures, target dose). Comparison participants will be asked about the acceptability of not getting the Bootle Blast program right away.
Monitoring Coach Logbook | Weeks 0-12 (Experimental Group), Weeks 12-24 (Waitlist Comparison Group).
  Documentation of weekly coach contacts (duration, content type, informational/motivational support) to assess feasibility and perceived value of coach involvement.
Technical Assistance Requests | Weeks 0-12 (Experimental Group), Weeks 12-24 (Waitlist Comparison Group).
  Frequency and nature of technical support inquiries related to Bootle Blast equipment setup, functionality, and home use.
Semi-Structured Interviews | Week 12 (Experimental Group), Week 24 (Waitlist Comparison Group).
  Qualitative interviews exploring enablers and barriers to engagement, motivational factors, and experience with the intervention. Conducted separately with children and caregivers.
Engagement (PRIME-C and PRIME-P) | Weeks 1, 6, and 12 of each participant's Bootle Blast intervention period.
  Parent- and child-reported engagement using the Pediatric Rehabilitation Intervention Measure of Engagement (affective, behavioral, cognitive components).
In-Game Engagement Prompts | Weekly during Bootle Blast intervention.
  Child-reported ratings of enjoyment, challenge, and effort through weekly in-game prompts.

SECONDARY OUTCOMES:
Quality of Upper Extremity Skills Test (QUEST) | Baseline, 12 weeks, 24 weeks.
  Unimanual domain scores assessing dissociated movement, grasp, weight bearing, and protective extension.
Grip Strength (Modified Sphygmomanometer) | Baseline, 12 weeks, 24 weeks.
  Grip strength of the hemiplegic hand as an indicator of selective motor control.
Active Range of Motion (aROM) | Baseline, 12 weeks, 24 weeks.
  Active range of motion of wrist, elbow, and shoulder on the hemiplegic side measured using a manual goniometer.
Box and Block Test (BBT) | Baseline, 12 weeks, 24 weeks.
  Manual dexterity measured as the number of blocks transferred in one minute for each hand.
Assisting Hand Assessment (AHA) | Baseline, 12 weeks, 24 weeks.
  Evaluates spontaneous use and effectiveness of the impaired hand during bimanual activities.
Shriners Hospital Upper Extremity Evaluation - Spontaneous Functional Analysis (SHUEE-SFA) | Baseline, 12 weeks, 24 weeks.
  The 15 min SHUEE is designed for children with spastic hemiplegic CP aged 3 to 18 years. This measure was designed by the Shriners Hospital for Children to evaluate functional and spontaneous ability, and dynamic segmental alignment of the upper limb of children with hemiplegic CP. The SHUEE includes the assessment of active and passive range of motion, tone, performance of activities of daily living (client reported) and evaluation of 16 activities using the hand and arm. The assessment is videorecorded and scored at a later time. Of note, in this study, sections of the SHUEE (aROM, performance of activities of daily living) will be excluded as they will be captured separately. The 16 hand and arm activities are evaluated based on the dynamic segmental alignment (DSA) and the spontaneous functional analysis (SFA) of the involved UL. The scoring uses a numerical scale from 0-5 for the SFA, and 0-3 for the DSA, where 0 is the lowest / less functional score.
Canadian Occupational Performance Measure (COPM) | Baseline, 12 weeks, 24 weeks.
  Three child/family-identified goals related to activities of everyday living (e.g. self-care, leisure) that they hope to improve on. Participants then rate their performance and satisfaction for each goal/challenge area on a scale from 1 to 10 (low to high). Average scores for performance and satisfaction are calculated across the goals. The COPM is extensively used with children with CP in the target age range and with success in the research team's pilot work. It has good validity, responsiveness, reliability, and ability to track change over time. A change of 2 points on either the performance or satisfaction scale is considered clinically significant.
Performance Quality Rating Scale (PQRS) | Biweekly throughout the 24-week study.
  Rater-scored (1-10) analysis of caregiver-recorded videos of child performing COPM-related tasks, assessing accuracy, timeliness, safety, and overall quality. Assessors will be trained on practice videos to establish consistent scoring practices. Assessors will be blinded to the time point at which the video recording was collected.
Children's Hand-use Experience Questionnaire (CHEQ) | Baseline, 12 weeks, 24 weeks.
  Caregiver-reported quality and effectiveness of the child's use of the affected hand in 29 bimanual activities.
Inertial Sensor Activity Counts (Optional) | Baseline, Week 12 and Week 24; Pre- and post-intervention (5 consecutive days each period).
  Wrist-worn inertial sensor data assessing continuous daily hand/arm activity in a child's natural context, including the ratio of non-dominant to dominant arm activity. As long as they are acceptable and do not interfere with the assessments, children will be asked to wear inertial sensors on their wrists during the assessment sessions. Additionally, for those who are willing and subject to availability of sensors, children will be asked to wear the inertial sensors for 5 consecutive days (at least 6 hours per day) at home pre- and post-intervention.
Bootle Blast Computer Logs | Weeks 0-12 (Experimental Group), Weeks 12-24 (Waitlist Comparison Group).
  Computer logs will be used as a measure of adherence to the Bootle Blast intervention. Every time the computer is turned on to play, a video game log is automatically generated. These logs will record details for each play session providing information about active play time, game performance and progress. The game logs active (i.e., minutes spent actively engaging in therapeutic movements) and passive play time (e.g., time spent navigating menus). Additional data recorded in game logs include game scores, games played, and rewards collected, as well as skeletal data and video footage of game play if participants have consented to the latter. Data will be securely uploaded and saved into the cloud (Cloud Storage for Firebase & Cloud Firestore by Google, servers in Montreal, Canada).
Child Mood, Energy, and Pain Ratings | Baseline, 12 weeks, 24 weeks.
  Self-reported ratings of mood, fatigue (battery scale), and pain (Wong-Baker FACES) at each clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital, Bloorview Research Institute; Virginia Wright, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital, Bloorview Research Institute
Locations (3):
- Canada (3):
  - Grandview Kids, Ajax, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No